CLINICAL TRIAL: NCT03247504
Title: Adherence to Opioids in Oncology Out Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0436
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Cancer Out Patients With Opioids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer pain is undertreated despite a good access to opioids in France. Although many factors are involved, the barriers related to the patient (and his family) are often reported .the reluctance of the patient or the family to take the prescribed medication is linked to misconceptions about the opioids , cultural barriers; or the lack of explanations provided by the physician. Some patients can have undiagnosed slight cognitive impairment .The situation is now more complicated as appear on the market the new form of opioids for the cancer breakthrough pain drug, adding one more opioid formulation in the prescription. The goal of the study is to measure the adherence to opioids in cancer out patients and the associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Cancer out patients with opioids by mouth prescription
* Prescription than more than 8 days

Exclusion Criteria:

* Patient not at home, but in nursing home or other setting were the treatment are given by medical staff
* Patient unable to answer at the questionnaire
* Opoids given Intravenous or other way than mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer out patients with opioids treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Rate of cancer out patients with a low adherence to the opioids treatment | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Soins Palliatifs Lyon-Sud, Pierre-Bénite, France